CLINICAL TRIAL: NCT06293417
Title: To Assess the Long-term Efficacy and Safety of Combined Therapy With Ezefeno Tab. in Patients With Dyslipidemia Who do Not Achieve Adequate Control of Non-HDL-C Levels Even With Moderate-intensity Monotherapy
Brief Title: To Assess With Ezefeno Tab. in Patients With Dyslipidemia and T2DM
Acronym: ENSEMBLE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Korea University Anam Hospital (Other)
Responsible Party: Principal Investigator, Sin Gon Kim, professor, Korea University Anam Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HT-EF-01
Record Dates: First submitted 2024-02-19; First posted 2024-03-05 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: T2DM (Type 2 Diabetes Mellitus); Dyslipidemias
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Dyslipidemias | interventions — Ezetimibe; Fenofibrate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Ezetimibe/fenofibrate (Ezefeno) and moderate-intensity statin
  Interventions: Drug: Ezetimibe/fenofibrate (Ezefeno) and moderate-intensity statin
- Control group (Active Comparator): Dose escalation of moderate-intensity statin
  Interventions: Drug: Dose escalation of moderate-intensity statin

INTERVENTIONS:
Drug: Ezetimibe/fenofibrate (Ezefeno) and moderate-intensity statin — Treatment group
  Arms: Treatment group
Drug: Dose escalation of moderate-intensity statin — Control group
  Arms: Control group

SUMMARY:
The goal of this Randomized controlled trials is to assess in the long term efficacy and safety of ezefeno. The primary endpoint are:

* major adverse cardiovascular events within 48 months of the trial duration
* microvascular events within 48 months of the trial duration

DETAILED DESCRIPTION:
A prospective, randomized, open-label, parallel, multicenter, active-drug-controlled clinical trial to assess the long-term efficacy and safety of Combined Therapy with Ezefeno Tab. in patients with dyslipidemia who do not achieve adequate control of Non-HDL-C levels even with Moderate-intensity monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes diagnosed by American Diabetes Association criteria
* Age ≥ 19 years
* Non-HDL-C ≥100 mg/dL, TG ≥200, <500 mg/dL on moderate-intensity statins
* with cardiovascular risk factor

Exclusion Criteria:

* Pregnant or breastfeeding women
* Uncontrolled hyperglycemia(more than 12.0% for Subject treated with anti-diabetic treatment.)
* Patient with myopathy and rhabdomyolysis
* AST/ALT more than 3 ULN
* Clinical evidence of genetic disorders such as galactose intolerance, Lapp lactose deficiency, and/or glucose-galactose malabsorption

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3958 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
major adverse cardiovascular events and diabetic microvascular events for 48 months | 48month from baseline
  major adverse cardiovascular events and diabetic microvascular events for 48 months

SECONDARY OUTCOMES:
proportion of patients achieving Non-HDL-C less than 100mg/dL | 48month from baseline
  proportion of patients achieving Non-HDL-C less than 100mg/dL
proportion of patients achieving LDL less than 70mg/dL | 48month from baseline
  proportion of patients achieving LDL less than 70mg/dL
change in Non-HDL-C at 48month from baseline | 48month from baseline
  change in Non-HDL-C at 48month from baseline
change in LDL at 48month from baseline | 48month from baseline
  change in LDL at 48month from baseline
change in HDL-C at 48month from baseline | 48month from baseline
  change in HDL-C at 48month from baseline
change in TG at 48month from baseline | 48month from baseline
  change in TG at 48month from baseline
change in LDL-C/HDL-C ratio at 48month from baseline | 48month from baseline
  change in LDL-C/HDL-C ratio at 48month from baseline
change in TC/HDL-C ratio at 48month from baseline | 48month from baseline
  change in TC/HDL-C ratio at 48month from baseline

CONTACTS AND LOCATIONS:
Overall Officials: SIN-GON KIM, Principal Investigator — Korea University Anam Hospital
Locations (1):
- Korea University Anam Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided